CLINICAL TRIAL: NCT06124989
Title: A Novel Machine Learning Model for the Prediction of Relapse of Acute Biliary Pancreatitis (Machine learnINg for the rElapse Risk eValuation in Acute Biliary Pancreatitis - MINERVA)
Brief Title: Machine learnINg for the rElapse Risk eValuation in Acute Biliary Pancreatitis.
Acronym: MINERVA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Università di Napoli Federico II (Unknown); Università della Campania Luigi Vanvitelli (Unknown)
Responsible Party: Principal Investigator, Mauro Podda, Prof., University of Cagliari
Other Study IDs: MINERVA_1
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Pancreatitis; Pancreatitis Due to Gallstones; Pancreatitis Biliary; Pancreatitis Relapsing
Keywords: Machine Learning, Prediction Model
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MINERVA Machine Learning model — The MINERVA score for the prediction of the risk of relapse of acute pancreatitis in patients who did not undergo early cholecystectomy after the first episode of acute biliary pancreatitis will be grounded upon a Machine Learning model that takes into account patients' demographic, clinical, and laboratory variables that can be easily collected and recorded at index patient admission.

SUMMARY:
The MINERVA (Machine learnINg for the rElapse Risk eValuation in Acute biliary pancreatitis) project stems from the need in the clinical practice of taking an operational decision in patients that are admitted to the hospital with a diagnosis of acute biliary pancreatitis. In particular, the MINERVA prospective cohort study aims to develop a predictive score that allows to assess the risk of hospital readmission for patients diagnosed with mild biliary acute pancreatitis using Machine Learning and artificial intelligence.

The objectives of the MINERVA study are to:

1. Propose a novel methodology for the assessment of the risk of relapse in patients with mild biliary acute pancreatitis who did not undergo early cholecystectomy (within 3 to 7 days from hospital admission);
2. Propose a Machine Learning predictive model using a Deep Learning architecture applied to easily collectable data;
3. Validate the MINERVA score on an extensive, multicentric, prospective cohort;
4. Allow national and international clinicians, medical staff, researchers and the general audience to freely and easily access the MINERVA score computation and use it in their daily clinical practice.

The MINERVA score model will be developed on a retrospective cohort of patients (MANCTRA-1, already registered in ClinicalTrials.gov) and will be validated on a novel prospective multicentric cohort. After validation, the MINERVA score will be free and easy to compute instantly for all medical staff; it will be accessible at any time on the MINERVA website and web app, and will provide an immediate and reliable result that can be a clear indication for the best treatment pathway for the clinician and for the patient.

DETAILED DESCRIPTION:
Acute pancreatitis is the most common pancreatic disease, with a global incidence of 34 cases per 100,000 individuals. This disease counts more than 1.5 million new patients per year worldwide, with a mortality that approaches 1%. Mild biliary acute pancreatitis patients, when admitted to the hospital, can be treated with index, early cholecystectomy (within 3 to 7 days from the acute episode) or conservatively. While conservative treatment can be resolutive, up to 35% of these patients have a relapse within 30 days, and require emergency surgery in a significantly worse overall patient condition, reducing the chances of success. Other than that, relapse dramatically increases the chances of chronic pancreatitis, pancreatic cancer, postoperative complications and overall mortality. Relapse episodes have also an economic impact on healthcare facilities, as a second and longer hospital admission per patient increases the overall medical cost per patient by at least 100%. So far, however, there are no standardised methods to predict relapse of biliary acute pancreatitis in patients who did not undergo early cholecystectomy after the first episode of mild biliary acute pancreatitis.

The MINERVA (Machine learnINg for the rElapse Risk eValuation in Acute biliary pancreatitis) project stems from the need in the clinical practice of taking an operational decision in patients that are admitted to the hospital with a diagnosis of mild acute biliary pancreatitis.

The MINERVA project aims to reach the following objectives and results:

1. Propose a novel methodology for the assessment of the risk of relapse in patients with mild biliary acute pancreatitis who did not undergo early cholecystectomy after the first episode of mild biliary acute pancreatitis;
2. Propose a Machine Learning predictive model using a Deep Learning architecture applied to data easy to collect from patients;
3. Validate the MINERVA score on an extensive, multicentric, prospective cohort;
4. Allow national and international clinicians, medical staff, researchers and the general audience to freely and easily access the MINERVA score computation and use it in their daily clinical practice.

The MINERVA score will provide the clinicians with a validated and standardized assessment of relapse risk that takes into account the personal history, demographic data and laboratory characteristics of each patient. The MINERVA score will be free and easy to compute instantly for all medical staff; it will be accessible at any time on the MINERVA website and web app, and will provide an immediate and reliable result that can be a clear indication for the best treatment pathway for the clinician and for the patient.

The MINERVA score model will be developed on a retrospective cohort of patients (MANCTRA-1, already registered in ClinicalTrials.gov) and will be validated on a novel prospective multicentric cohort.

Retrospective cohort The model development and initial training will be performed on a retrospective cohort of patients (n=692) collected during a preliminary multicentric study, the MANCTRA-1 study (approved by the Ethics Committee of the University of Cagliari Hospital, MANCTRA-1 - NCT04747990, Prot. PG/2021/7108) conducted by the PI (Dr. Mauro Podda) and the University of Cagliari local responsible of the MINERVA project.

Prospective cohort A total of 430 patients will be recruited in the prospective cohort of the MINERVA study.

Methods The MINERVA score will be grounded on a Machine Learning model that will be developed and trained on a retrospective cohort and validated on a prospective cohort of patients.

All model variables will be processed with kernel Principal Component Analysis (kPCA).

The Convex Hull of the scatterplot of the main components will be computed and the smallest rectangle will be extracted. The rectangle will be transformed into a 2d image with a fixed resolution using feature averaging and normalization.

The model will be developed at the University of Naples Federico II by Dr. Daniela Pacella with the Machine Learning expertise and supervision.

To prevent overfitting, the dataset will be split into training set, test set and validation set. Additionally, k-fold cross-validation will be used. The performance of the MINERVA model will be evaluated using the most adopted measures of accuracy, such as precision, recall and AUC (Area Under the ROC Curve). Additionally, its performance will be compared with that achieved using traditional machine learning methods (SVM, ANN). Missing data will be handled with imputation methods.

Variables Age (Years) Sex (Male:Female) Previous episodes of biliary pancreatitis (Yes; No) Admitting speciality (HepatoPancreatoBiliary surgery, General surgery, Internal medicine, Gastroenterology) Body mass index -BMI- (Kg/m2) Clinical history of diabetes (No diabetes; Yes with organ dysfunction; Yes without organ dysfunction) Clinical history of chronic pulmonary disease (Yes; No) Clinical history of hypertension (Yes; No) Clinical history of atrial fibrillation (Yes; No) Clinical history of ischemic heart disease (Yes; No) Clinical history of chronic kidney disease (No; Yes under medications; Yes in permanent renal replacement therapy or in preparation for it) Clinical history of of diseases of the hematopoietic system (Yes; No) Patient on immunosuppressive medications on hospital admission (Yes; No) White Blood Cells -WBC- (cells/mm3) Neutrophils (cells/mm3) Platelets (Plt/mm3) INR (International Normalized Ratio) C-reactive protein -CRP- (mg/L) Aspartate aminotransferase -AST- (U/L) Alanine aminotransferase -ALT- (U/L) Total bilirubin (mg/dL) Conjugated bilirubin (mg/dL) Gamma-glutamil-transpeptidase -GGT- (U/L) Serum amylase (U/L) Serum lipase (U/L) Lactate DeHydrogenase -LDH- (U/L) Choledocholithiasis (Yes; Yes with common bile duct obstruction; No) Cholangitis (Yes; No) ERCP with sphincterotomy (Yes within 24h from hospital admission; Yes within 24-48h from hospital admission; Yes within 48-72h from hospital admission; No) Acute biliary pancreatitis relapse at 30-day, 60-day, 90-day, 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Clinical diagnosis of mild biliary acute pancreatitis (according to the Revised Atlanta Classification)
* Not submitted to cholecystectomy or ERCP/ES (Endoscopic Retrograde CholangioPancreatography/Endoscopic Sphyncterotomy) during the same hospital admission

Exclusion Criteria:

* Acute pancreatitis of etiology other than gallstones;
* Moderately-severe pancreatitis;
* Severe pancreatitis;
* Presence of pancreatic necrosis;
* Pregnant patients;
* Patients not able to sign the informed consent to take part in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old), of both sexes, admitted to the participating centers (surgical departments and/or gastroenterology departments and/or internal medicine departments) with a clinical diagnosis of mild biliary acute pancreatitis (according to the Revised Atlanta Classification), confirmed by at least an ultrasound scan, and not submitted to cholecystectomy or ERCP/ES (Endoscopic Retrograde CholangioPancreatography/Endoscopic Sphyncterotomy) during the same hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with recurrence of biliary acute pancreatitis. | 30-day, 60-day, 90-day, 1-year
  The number of patients with recurrence of biliary acute pancreatitis: prediction of risk relapse of acute biliary pancreatitis in patients after a first episode of mild biliary acute pancreatitis (according to the 2012 Revised Atlanta Classification) not submitted to early (within three to seven days from the acute episode) cholecystectomy. This outcome will be reached by the development and validation of a novel risk score.

SECONDARY OUTCOMES:
Accuracy of the MINERVA model. | 30-day, 60-day, 90-day, 1-year
  Accuracy, sensibility, and specificity (AUC, area under the ROC curve) of the MINERVA Machine Learning model compared with other traditional machine learning models previously adopted in literature (such as ANN and SVM) and with statistical models (such as multiple regression).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Podda, MD, Study Chair — University of Cagliari, Department of Surgical Science
Locations (1):
- University of Cagliari, Emergency Surgery Department, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Ahmed Ali U, Issa Y, Hagenaars JC, Bakker OJ, van Goor H, Nieuwenhuijs VB, Bollen TL, van Ramshorst B, Witteman BJ, Brink MA, Schaapherder AF, Dejong CH, Spanier BW, Heisterkamp J, van der Harst E, van Eijck CH, Besselink MG, Gooszen HG, van Santvoort HC, Boermeester MA; Dutch Pancreatitis Study Group. Risk of Recurrent Pancreatitis and Progression to Chronic Pancreatitis After a First Episode of Acute Pancreatitis. Clin Gastroenterol Hepatol. 2016 May;14(5):738-46. doi: 10.1016/j.cgh.2015.12.040. Epub 2016 Jan 6. PMID 26772149
- [Background] Bagepally BS, Haridoss M, Sasidharan A, Jagadeesh KV, Oswal NK. Systematic review and meta-analysis of gallstone disease treatment outcomes in early cholecystectomy versus conservative management/delayed cholecystectomy. BMJ Open Gastroenterol. 2021 Jul;8(1):e000675. doi: 10.1136/bmjgast-2021-000675. PMID 34261757
- [Background] Chen Y, Chen TW, Wu CQ, Lin Q, Hu R, Xie CL, Zuo HD, Wu JL, Mu QW, Fu QS, Yang GQ, Zhang XM. Radiomics model of contrast-enhanced computed tomography for predicting the recurrence of acute pancreatitis. Eur Radiol. 2019 Aug;29(8):4408-4417. doi: 10.1007/s00330-018-5824-1. Epub 2018 Nov 9. PMID 30413966
- [Background] Cho JH, Jeong YH, Kim KH, Kim TN. Risk factors of recurrent pancreatitis after first acute pancreatitis attack: a retrospective cohort study. Scand J Gastroenterol. 2020 Jan;55(1):90-94. doi: 10.1080/00365521.2019.1699598. Epub 2019 Dec 10. PMID 31822144
- [Background] da Costa DW, Bouwense SA, Schepers NJ, Besselink MG, van Santvoort HC, van Brunschot S, Bakker OJ, Bollen TL, Dejong CH, van Goor H, Boermeester MA, Bruno MJ, van Eijck CH, Timmer R, Weusten BL, Consten EC, Brink MA, Spanier BWM, Bilgen EJS, Nieuwenhuijs VB, Hofker HS, Rosman C, Voorburg AM, Bosscha K, van Duijvendijk P, Gerritsen JJ, Heisterkamp J, de Hingh IH, Witteman BJ, Kruyt PM, Scheepers JJ, Molenaar IQ, Schaapherder AF, Manusama ER, van der Waaij LA, van Unen J, Dijkgraaf MG, van Ramshorst B, Gooszen HG, Boerma D; Dutch Pancreatitis Study Group. Same-admission versus interval cholecystectomy for mild gallstone pancreatitis (PONCHO): a multicentre randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1261-1268. doi: 10.1016/S0140-6736(15)00274-3. PMID 26460661
- [Background] Ding N, Guo C, Li C, Zhou Y, Chai X. An Artificial Neural Networks Model for Early Predicting In-Hospital Mortality in Acute Pancreatitis in MIMIC-III. Biomed Res Int. 2021 Jan 28;2021:6638919. doi: 10.1155/2021/6638919. eCollection 2021. PMID 33575333
- [Background] Gurusamy KS, Nagendran M, Davidson BR. Early versus delayed laparoscopic cholecystectomy for acute gallstone pancreatitis. Cochrane Database Syst Rev. 2013 Sep 2;2013(9):CD010326. doi: 10.1002/14651858.CD010326.pub2. PMID 23996398
- [Background] Hong WD, Chen XR, Jin SQ, Huang QK, Zhu QH, Pan JY. Use of an artificial neural network to predict persistent organ failure in patients with acute pancreatitis. Clinics (Sao Paulo). 2013 Jan;68(1):27-31. doi: 10.6061/clinics/2013(01)rc01. No abstract available. PMID 23420153
- [Background] Mashayekhi R, Parekh VS, Faghih M, Singh VK, Jacobs MA, Zaheer A. Radiomic features of the pancreas on CT imaging accurately differentiate functional abdominal pain, recurrent acute pancreatitis, and chronic pancreatitis. Eur J Radiol. 2020 Feb;123:108778. doi: 10.1016/j.ejrad.2019.108778. Epub 2019 Dec 11. PMID 31846864
- [Background] Hu X, Yang B, Li J, Bai X, Li S, Liu H, Zhang H, Zeng F. Individualized Prediction of Acute Pancreatitis Recurrence Using a Nomogram. Pancreas. 2021 Jul 1;50(6):873-878. doi: 10.1097/MPA.0000000000001839. PMID 34347724
- [Background] Loozen CS, Oor JE, van Ramshorst B, van Santvoort HC, Boerma D. Conservative treatment of acute cholecystitis: a systematic review and pooled analysis. Surg Endosc. 2017 Feb;31(2):504-515. doi: 10.1007/s00464-016-5011-x. Epub 2016 Jun 17. PMID 27317033
- [Background] Mador BD, Panton ON, Hameed SM. Early versus delayed cholecystectomy following endoscopic sphincterotomy for mild biliary pancreatitis. Surg Endosc. 2014 Dec;28(12):3337-42. doi: 10.1007/s00464-014-3621-8. Epub 2014 Jun 25. PMID 24962855
- [Background] Nebiker CA, Frey DM, Hamel CT, Oertli D, Kettelhack C. Early versus delayed cholecystectomy in patients with biliary acute pancreatitis. Surgery. 2009 Mar;145(3):260-4. doi: 10.1016/j.surg.2008.10.012. Epub 2009 Feb 1. PMID 19231577
- [Background] Riquelme F, Marinkovic B, Salazar M, Martinez W, Catan F, Uribe-Echevarria S, Puelma F, Munoz J, Canals A, Astudillo C, Uribe M. Early laparoscopic cholecystectomy reduces hospital stay in mild gallstone pancreatitis. A randomized controlled trial. HPB (Oxford). 2020 Jan;22(1):26-33. doi: 10.1016/j.hpb.2019.05.013. Epub 2019 Jun 22. PMID 31235428
- [Background] Sankaran SJ, Xiao AY, Wu LM, Windsor JA, Forsmark CE, Petrov MS. Frequency of progression from acute to chronic pancreatitis and risk factors: a meta-analysis. Gastroenterology. 2015 Nov;149(6):1490-1500.e1. doi: 10.1053/j.gastro.2015.07.066. Epub 2015 Aug 20. PMID 26299411
- [Background] Schmidt M, Sondenaa K, Vetrhus M, Berhane T, Eide GE. A randomized controlled study of uncomplicated gallstone disease with a 14-year follow-up showed that operation was the preferred treatment. Dig Surg. 2011;28(4):270-6. doi: 10.1159/000329464. Epub 2011 Jul 9. PMID 21757915
- [Background] Sharma A, Vans E, Shigemizu D, Boroevich KA, Tsunoda T. DeepInsight: A methodology to transform a non-image data to an image for convolution neural network architecture. Sci Rep. 2019 Aug 6;9(1):11399. doi: 10.1038/s41598-019-47765-6. PMID 31388036
- [Background] Stevens CL, Abbas SM, Watters DA. How Does Cholecystectomy Influence Recurrence of Idiopathic Acute Pancreatitis? J Gastrointest Surg. 2016 Dec;20(12):1997-2001. doi: 10.1007/s11605-016-3269-x. Epub 2016 Sep 23. PMID 27663692
- [Background] Umans DS, Hallensleben ND, Verdonk RC, Bouwense SAW, Fockens P, van Santvoort HC, Voermans RP, Besselink MG, Bruno MJ, van Hooft JE; Dutch Pancreatitis Study Group. Recurrence of idiopathic acute pancreatitis after cholecystectomy: systematic review and meta-analysis. Br J Surg. 2020 Feb;107(3):191-199. doi: 10.1002/bjs.11429. Epub 2019 Dec 25. PMID 31875953
- [Background] Werner J, Hartwig W, Uhl W, Muller C, Buchler MW. Useful markers for predicting severity and monitoring progression of acute pancreatitis. Pancreatology. 2003;3(2):115-27. doi: 10.1159/000070079. PMID 12748420
- [Background] Yamashita R, Nishio M, Do RKG, Togashi K. Convolutional neural networks: an overview and application in radiology. Insights Imaging. 2018 Aug;9(4):611-629. doi: 10.1007/s13244-018-0639-9. Epub 2018 Jun 22. PMID 29934920
- [Background] Yuan X, Xu B, Wong M, Chen Y, Tang Y, Deng L, Tang D. The safety, feasibility, and cost-effectiveness of early laparoscopic cholecystectomy for patients with mild acute biliary pancreatitis: A meta-analysis. Surgeon. 2021 Oct;19(5):287-296. doi: 10.1016/j.surge.2020.06.014. Epub 2020 Jul 22. PMID 32709425
- [Background] Zhou Y, Ge YT, Shi XL, Wu KY, Chen WW, Ding YB, Xiao WM, Wang D, Lu GT, Hu LH. Machine learning predictive models for acute pancreatitis: A systematic review. Int J Med Inform. 2022 Jan;157:104641. doi: 10.1016/j.ijmedinf.2021.104641. Epub 2021 Nov 10. PMID 34785488
- [Derived] Podda M, Pisanu A, Pellino G, De Simone A, Selvaggi L, Murzi V, Locci E, Rottoli M, Calini G, Cardelli S, Catena F, Vallicelli C, Bova R, Vigutto G, D'Acapito F, Ercolani G, Solaini L, Biloslavo A, Germani P, Colutta C, Occhionorelli S, Lacavalla D, Sibilla MG, Olmi S, Uccelli M, Oldani A, Giordano A, Guagni T, Perini D, Pata F, Nardo B, Paglione D, Franco G, Donadon M, Di Martino M, Bruzzese D, Pacella D. Machine learning for the rElapse risk eValuation in acute biliary pancreatitis: The deep learning MINERVA study protocol. World J Emerg Surg. 2025 Mar 3;20(1):17. doi: 10.1186/s13017-025-00594-7. PMID 40033414